CLINICAL TRIAL: NCT06657742
Title: Validity and Reliability of the Turkish Version of the Spinal Cord Independence Measure Self-Report
Brief Title: Validity and Reliability of SCIM-SR
Status: Completed | Type: Observational
Sponsor: Istanbul Physical Medicine Rehabilitation Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Yelda Soluk Özdemir, Principle investigator, Istanbul Physical Medicine Rehabilitation Training and Research Hospital
Other Study IDs: 2023/385
Record Dates: First submitted 2024-10-22; First posted 2024-10-24 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: SCIM-SR — SCIM-SR was a self-reported scale that evaluated the independence of patients.

SUMMARY:
To determine the validity and reliability of SCIM-SR, patients will fill out SCIM 3 and SR.

DETAILED DESCRIPTION:
To determine the validity and reliability of SCIM-SR, patients will fill out SCIM 3 and SR. scım-sr Turkish form has been created. Patients with spinal cord injuries who applied to our physical therapy clinic filled out the form twice.

ELIGIBILITY:
Inclusion Criteria:

* SCI >1 month
* 18-70 years
* agree to participate
* give written consent

Exclusion Criteria:

* not read Turkish,
* not write Turkish,
* cognitive problems

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: -SCI patients between the ages of 18-70 and at least 1 month after their injury
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2023-10-16 (Actual); Primary Completion 2024-06-16 (Actual); Study Completion 2024-07-16 (Actual)

PRIMARY OUTCOMES:
SCIM-SR | baseline
  scım-sr was a self-reported scale that evaluated the independence of patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Cansın Medin Ceylan, Istanbul, None Selected, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No